CLINICAL TRIAL: NCT05681962
Title: Practice of Oxygenation and Respiratory Support During Fiberoptic Bronchoscopy: the Oxy-FOB STUDY
Brief Title: Practice of Oxygenation and Respiratory Support During Fiberoptic Bronchoscopy
Status: Recruiting | Type: Observational
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Director of the Intensive Care and Anesthesia Department, University Magna Graecia
Other Study IDs: OxyFOB study
Record Dates: First submitted 2023-01-03; First posted 2023-01-12 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Acute Respiratory Failure; Pneumonia; Lung Cancer; Fibrosis Lung; Interstitial Lung Disease
Keywords: Bronchoscopy
MeSH Terms: conditions — Pneumonia; Lung Neoplasms; Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Standard Oxygen Therapy (SOT): Patients receiving low oxygen flow administration through nasal prongs, oxygen mask with or without reservoir, and Venturi mask.
  Interventions: Diagnostic Test: Bronchoscopy
- High Flow oxygen through Nasal Cannula (HFNC): Administration of high flows (up to 60 L/min) of air/oxygen admixtures, heated (at temperatures ranging from 31 to 37°C) and fully humidified (up to 44 mg H2O/L), providing an inspired oxygen fraction ranging from 21 to 100%
  Interventions: Diagnostic Test: Bronchoscopy
- Continuous Positive Airway Pressure (CPAP): application of positive end-expiratory pressure (PEEP) throughout the whole respiratory cycle by means of interfaces such as mask or helmet
  Interventions: Diagnostic Test: Bronchoscopy
- Non-Invasive Ventilation (NIV): application of a PEEP by means of a mask or helmet, with an inspiratory pressure support triggered by the patient and delivered by a ventilator and through interfaces such as mask or helmet
  Interventions: Diagnostic Test: Bronchoscopy
- Invasive Mechanical Ventilation (iMV): application of a ventilatory assistance in controlled or partial assisted modalities through an endotracheal or tracheostomy tube
  Interventions: Diagnostic Test: Bronchoscopy

INTERVENTIONS:
Diagnostic Test: Bronchoscopy — Patients will undergo to the bronchial endoscopy procedure required for their clinical condition: toilet bronchoscopy (for secretions, blood, mucus plugs removal), broncho-aspirate (BAS), bronchoalveolar lavage (BAL), brushing for cytology, biopsy, endobronchial ultrasound (EBUS).

SUMMARY:
The current practice of oxygenation and/or ventilation supports in patients undergoing Fiberoptic Bronchoscopy is very heterogeneous among studies published in the literature; in addition, clear outcomes advantages of one strategy over another currently lack.

The goal of this observational study is to describe the current practice of oxygenation and/or ventilation supports in patients undergoing Fiberoptic Bronchoscopy (FOB), stratified by baseline respiratory condition, co-morbidities, type of procedure and hospital settings.

Investigators will enroll all adult patients undergoing any fiberoptic bronchoscopy in any clinical settings (from outpatients to critically ill patients). No specific exclusion criteria are indicated for enrollment in this study.

Investigators will record the following data:

* Patient's baseline data.
* Type of FOB procedure: toilet bronchoscopy (for secretions, blood, mucus plugs removal), broncho-aspirate (BAS), bronchoalveolar lavage (BAL), brushing for cytology, biopsy, endobronchial ultrasound (EBUS). The type and size of bronchoscope (with or without an internal/external camera) and the time of the procedure will be also recorded.
* Type of supportive strategy: no support, Standard Oxygen Therapy, High Flow Nasal Cannula, Continuous Positive Airway Pressure and or non invasive ventilation trough mask or helmet, invasive mechanical ventilation.
* Sedation
* Intra-procedural vital parameters
* Occurrence of adverse events: desaturation (i.e. SpO2< 90% for at least 10 seconds), severe desaturation (i.e. SpO2< 80%), need for procedure interruption, hypotensive (systolic blood pressure <90 mmHg) or hypertensive (systolic blood pressure >140 mmHg) events, new onset of cardiac arrhythmias (specify the rhythm) or myocardial ischemia or electrocardiographic ST-alterations, neurological events (i.e. severe sensorium depression, psychomotor agitation).
* Post-procedural vital parameters (15 minutes after the procedure).
* Clinical outcomes: need for support escalation, need for admission to ward (for outpatient) or ICU (for outpatients and ward-admitted patient).

ELIGIBILITY:
Inclusion Criteria:

* Need for any procedure with flexible FOB
* Either outpatients in dedicated ambulatories, and admitted to any hospital ward or Intensive Care Unit (ICU)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include all adult patients requiring a flexible bronchoscopy for diagnostic or procedural reasons from all possible settings (from outpatients in dedicated ambulatories to patients admitted in any hospital ward or Intensive Care Unit)
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Type of oxygenation strategy adopted | Through the endoscopy completion, an average of 30 minutes
  The type of oxygenation strategy (standard oxygen therapy, high flow nasal cannula, continuous positive airway pressure, non invasive ventilation or invasive mechanical ventilation) adopted during the bronchoscopy will be recorded.

SECONDARY OUTCOMES:
Type of sedation strategy adopted | Through the endoscopy completion, an average of 30 minutes
  The type of sedation strategy (topical anesthesia, midazolam, propofol, remifentanil, fentanyl, dexmedetomidine, neuromuscular blocking agents) adopted during the bronchoscopy will be recorded.
Lowest peripheral oxygen saturation | Through the endoscopy completion, an average of 30 minutes
  The lowest peripheral oxygen saturation recorded during the procedure
Lowest heart rate | Through the endoscopy completion, an average of 30 minutes
  The lowest heart rate recorded during the procedure
Highest heart rate | Through the endoscopy completion, an average of 30 minutes
  The highest heart rate recorded during the procedure
Lowest systolic blood pressure | Through the endoscopy completion, an average of 30 minutes
  The lowest systolic blood pressure recorded during the procedure
Highest systolic blood pressure | Through the endoscopy completion, an average of 30 minutes
  The highest systolic blood pressure recorded during the procedure
Duration of the procedure | From the beginning to the end of the endoscopy procedure
  The time duration of the procedure in minutes, from the beginning to the end of the endoscopy procedure
Desaturation events | Through the endoscopy completion, an average of 30 minutes
  Occurrence of peripheral oxygen saturation < 90% for at least 10 seconds
Severe desaturation events | Through the endoscopy completion, an average of 30 minutes
  Occurrence of peripheral oxygen saturation < 80%
Hypotensive events | Through the endoscopy completion, an average of 30 minutes
  Occurrence of systolic blood pressure <90 mmHg
Hypertensive events | Through the endoscopy completion, an average of 30 minutes
  Occurrence of systolic blood pressure >140 mmHg
Need for support escalation | Through the endoscopy completion, an average of 30 minutes
  Need to escalate the oxygenation/ventilation support from from standard oxygen therapy (lowest support) to High Flow Nasal Cannula, Continuous Positive Airway Pressure, Non Invasive Ventilation or invasive Mechanical Ventilation (highest grade of support)
Admission to ward or intensive care unit | At the end of the endoscopy completion, after an average of 30 minutes from study start
  Need for admission to ward or intensive care unit after the endoscopy completion

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be shared after study publication on a peer-reviewed journal in english language, on a reasonable request to the principal investigator
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After study publication on a peer-reviewed journal in english language
Access Criteria: On reasonable request to the Principal Investigator

REFERENCES:
- [Derived] Longhini F, Crimi C, Noto A, Pelaia C, Karakurt Z, Skoczynski S, Boleo-Tome JP, Winck JC, Esquinas AM, Melhorn J, Corneci D, Pobeha P, Bosco V, Garofalo E, Bruni A, Cammarota G, Todorova V, Puci MV, Sotgiu G, Kostikas K, Maggiore SM, De Robertis E, Ergan B, Landoni G, Simonte R, Nava S, Navalesi P, Scala R; OxyFOB study group. Practice of oxygenation and respiratory support during fibreoptic bronchoscopy: the OxyFOB study protocol. BMJ Open. 2025 Sep 2;15(9):e104747. doi: 10.1136/bmjopen-2025-104747. PMID 40897500